CLINICAL TRIAL: NCT04775173
Title: Efficacy and Safety of High- vs Low-Dose Sirolimus in Patients With Kaposiform Hemangioendothelioma: A Trial Protocol
Brief Title: Efficacy and Safety of Different Concentrations of Sirolimus in the Treatment of Kaposiform Hemangioendothelioma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Clinical Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-217
Record Dates: First submitted 2021-02-19; First posted 2021-03-01 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Kaposiform Hemangioendothelioma
Keywords: Kaposiform Hemangioendothelioma; Sirolimus; Efficacy; Safety
MeSH Terms: conditions — Kaposiform Hemangioendothelioma | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose of sirolimus (Experimental): Sirolimus The plasma trough concentration of sirolimus is maintained within the range of 5-8 ng/ml by adjusting sirolimus dose, for 1 year.
  Interventions: Drug: Sirolimus
- High dose of sirolimus (Active Comparator): Sirolimus The plasma trough concentration of sirolimus is maintained within the range of 10-15 ng/ml by adjusting sirolimus dose, for 1 year.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Use of different doses of the same drug
  Other Names: Rapamycin; Rapamune

SUMMARY:
The purpose of this study is to compare the efficacy and safety of different concentration gradients of sirolimus in the treatment of Kaposiform hemangioendothelioma.

DETAILED DESCRIPTION:
Kaposiform hemangioendothelioma (KHE) is a rare aggressive vascular neoplasm that occurs predominantly in infancy or early childhood, with an incidence of approximately 0.71/100,000. Currently, sirolimus is a promising treatment modality for KHE. Most scholars consider sirolimus blood concentration of 5-15 ng/ml to be an effective therapeutic concentration.

However, long-term higher dose sirolimus treatment can cause some common complications such as oral mucositis which affects the quality of life of the patient. Finer control of the plasma concentration of sirolimus may contribute to the efficacy of treatment and reduce the incidence of complications. Therefore, we conducted this study to see if low-dose sirolimus is beneficial to the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

Presenting a KHE with the following characteristics:

1. Male and female;
2. Between 0 and 14 years of age;
3. KHE diagnosis was confirmed by local investigators and by consensus of our multidisciplinary vascular anomaly group at the West China Hospital of Sichuan University based on:

   * Biopsy;
   * Compatible MRI findings;
   * History and clinical features.

   The multidisciplinary vascular anomaly group was a collaboration team that included vascular anomaly experts in pediatric surgery, plastic surgery, pediatric dermatology, pathology and radiology.
4. Without KMP, which was defined as a platelet count of less than 100×10^9/L, with consumptive coagulopathy and hypofibrinogenemia.
5. Patients were required to have adequate liver, renal and bone marrow function, and absence of active infection
6. Consent of parents (or the person with parental authority in families): signed and dated written informed consent.

Exclusion Criteria:

1. Patients contraindicated for the administration of sirolimus (e.g., those with an allergy to sirolimus or other rapamycin analog)
2. Exposure to chemotherapy, embolization, corticosteroids, propranolol, sclerotherapy or any other investigational agents within 1 weeks before enrolment on study;
3. Patients had a history of a major surgery within 2 weeks before enrollment;
4. Patients who have a history of treatment with sirolimus or other mTOR inhibitor;
5. Any known evidence of significant local or systemic uncontrolled infection, defined as receiving intravenous antibiotics at the time of enrollment;
6. Concurrent severe and/or uncontrolled medical diseases that could compromise participation in the study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe malnutrition, chronic liver or renal disease, active upper gastrointestinal tract ulceration).
7. Impairment of gastrointestinal function or chronic gastrointestinal disease that may significantly alter the absorption of sirolimus.
8. Patients with inadequate liver function:

   Total bilirubin higher than or equal to 1.5 × the upper limit of the normal (ULN) for age and alanine aminotransferase and aspartate aminotransferase higher than or equal to 2.5 × the ULN for age.
9. Patients with inadequate renal function:

   0-5 years of age maximum serum creatinine (mg/dL) of 0.8; 6-10 years of age maximum serum creatinine (mg/dL) of 1.0; 11-14 years of age maximum serum creatinine (mg/dL) of 1.2;
10. Adequate bone marrow function:

    Absolute neutrophil count lower than 1 × 109/L;
11. History of a malignancy within 5 years;
12. HIV infection or known immunodeficiency;
13. Indication for treatment with corticosteroids, vincristine, interferon-α, sirolimus, or tacrolimus for an indication other than IH;
14. Patients with an inability to participate in or follow-up during the study treatment and assessment plan;
15. Inability to give informed consent.

Ages: 1 Day to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
The proportion of patients achieving an objective response at month 12 | 12 months
  Objective response was defined as ≥20% reduction in KHE volume compared to that at baseline.

SECONDARY OUTCOMES:
lesion responses | 12 months
  The primary endpoint was classified as follow:
  * Complete involution: 100% resolution of the measured KHE;
  * Nearly complete involution was defined as decrease of ≥75% and <100%;
  * Partial involution was defined as decrease of ≥20% and <75%;
  * No change was defined as <20% increase and <20% decrease in the volumes of KHE lesions;
  * Further growth was defined as ≥20% increase in the volume of index KHE compared with the baseline volume measured. Lesion responses were overall lesion response rate and good lesion response rate.
  Overall lesion response comprised complete, nearly complete and partial involutions.
  Good lesion response comprised complete and nearly complete involutions.
Quality of life (QOL) in patients | 12 months
  Pediatric Quality of Life Inventory (PedsQLTM) 4.0 Genetic Core Infant Scales (<2 years) or Pediatric Quality of Life Inventory (PedsQLTM) 4.0 Genetic Core Scales (2-18 years) were used.
Disease sequelae | 12 months
  Disease sequelae (e.g., chronic pain, lymphedema and decreased ROM) were assessed by site investigators at month 12. The site investigators assessed patients' extremity swelling (if any), general physical activity and exercise levels. The diagnosis of lymphedema was based on physical examination (e.g., Stemmer's sign) and lymphoscintigraphic findings.
Frequency of adverse events | 12 months
  Frequency of adverse events (e.g. gastrointestinal disorders, blood and lymphatic system disorders, metabolic disorders or other abnormal laboratory results, skin disorders and general disorders, etc.) collected by investigator and reported by parents. All adverse events were collected and graded according to Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE v5.0). The causality of the adverse event was determined by the multidisciplinary staff and was classified as definitively not related, probably not related, possibly related, probably related, or definitively related. Any dose reductions, interruptions, or cessations enacted at the discretion of the investigators were recorded.
The changes of fibrinogen and D-dimer levels | 12 months
  Fibrinogen and D-dimer levels

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ji, MD, PhD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ji Y, Chen S, Yang K, Xia C, Li L. Kaposiform hemangioendothelioma: current knowledge and future perspectives. Orphanet J Rare Dis. 2020 Feb 3;15(1):39. doi: 10.1186/s13023-020-1320-1. PMID 32014025
- [Result] Ji Y, Chen S, Xiang B, Li K, Xu Z, Yao W, Lu G, Liu X, Xia C, Wang Q, Li Y, Wang C, Yang K, Yang G, Tang X, Xu T, Wu H. Sirolimus for the treatment of progressive kaposiform hemangioendothelioma: A multicenter retrospective study. Int J Cancer. 2017 Aug 15;141(4):848-855. doi: 10.1002/ijc.30775. Epub 2017 May 26. PMID 28486787
- [Result] Zhang G, Chen H, Gao Y, Liu Y, Wang J, Liu XY. Sirolimus for treatment of Kaposiform haemangioendothelioma with Kasabach-Merritt phenomenon: a retrospective cohort study. Br J Dermatol. 2018 May;178(5):1213-1214. doi: 10.1111/bjd.16400. Epub 2018 Mar 25. No abstract available. PMID 29388191
- [Result] Wang Z, Yao W, Sun H, Dong K, Ma Y, Chen L, Zheng S, Li K. Sirolimus therapy for kaposiform hemangioendothelioma with long-term follow-up. J Dermatol. 2019 Nov;46(11):956-961. doi: 10.1111/1346-8138.15076. Epub 2019 Sep 5. PMID 31489702
- [Result] Johnson AB, Richter GT. Vascular Anomalies. Clin Perinatol. 2018 Dec;45(4):737-749. doi: 10.1016/j.clp.2018.07.010. Epub 2018 Sep 18. PMID 30396415
- [Result] Adams DM, Ricci KW. Vascular Anomalies: Diagnosis of Complicated Anomalies and New Medical Treatment Options. Hematol Oncol Clin North Am. 2019 Jun;33(3):455-470. doi: 10.1016/j.hoc.2019.01.011. PMID 31030813
- [Result] Drolet BA, Trenor CC 3rd, Brandao LR, Chiu YE, Chun RH, Dasgupta R, Garzon MC, Hammill AM, Johnson CM, Tlougan B, Blei F, David M, Elluru R, Frieden IJ, Friedlander SF, Iacobas I, Jensen JN, King DM, Lee MT, Nelson S, Patel M, Pope E, Powell J, Seefeldt M, Siegel DH, Kelly M, Adams DM. Consensus-derived practice standards plan for complicated Kaposiform hemangioendothelioma. J Pediatr. 2013 Jul;163(1):285-91. doi: 10.1016/j.jpeds.2013.03.080. No abstract available. PMID 23796341